CLINICAL TRIAL: NCT00970190
Title: Olfactory Dysfunction of Rhinosinusitis - cAMP/Calcium Signaling Study
Brief Title: Olfactory Dysfunction of Rhinosinusitis - Cyclic Adenosine Monophosphate (cAMP)/Calcium Signaling Study
Acronym: cAMP
Status: Completed | Type: Observational
Sponsor: Greg Davis (Other)
Responsible Party: Sponsor-Investigator, Greg Davis, Assistant Professor, University of Washington
Organization: University of Washington (Other)
Other Study IDs: 36534-B
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Sinusitis
Keywords: sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples consist of discarded tissue resulting from the following clinical procedures: endoscopic sinus surgery for chronic sinusitis, endoscopic transnasal approach to the pituitary for pituitary tumor removal, endoscopic inferior turbinectomy or septoplasty for nasal congestion and endoscopic repair of CSF leaks. Samples will only be retained for 1 year post-surgery and then destroyed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study examines the biochemistry underlying human olfaction in both normal and diseased states.

The study aims are: 1. to determine the levels of cAMP in olfactory tissue from people with chronic rhinosinusitis and other nasal disorders. 2. to correlate preoperative olfactory function with cAMP levels from biopsied olfactory tissue. 3. to determine odorant and pheromone-mediated activation of cultured human olfactory sensory neurons using calcium imaging and 4. to determine odorant and pheromone-mediated activation of cultured human olfactory sensory neurons using "smell-chip" technology.

DETAILED DESCRIPTION:
Subject will be recruited from those scheduled to have endoscopic sinus surgery and similar procedures. This study uses the tissue that would normally be discarded during the surgical process. The tissue is cultured and frozen for purposes of the following testing:

odor detection and signal transduction, cyclic adenosine monophosphate and odor detection, the role of cAMP in olfactory dysfunction, and pheromone detection.

Only tissue that would normally be discarded during the course of the surgery will be used. The study does not interfere with or change any clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18 years old and over and scheduled for one of the following:

  * endoscopic sinus surgery for chronic sinusitis
  * endoscopic transnasal approach to the pituitary for pituitary tumor removal
  * endoscopic inferior turbinectomy or septoplasty for nasal congestion
  * endoscopic repair of cerebrospinal fluid (CSF) leaks

Exclusion Criteria:

* Subjects are excluded if they are unable to give informed consent or unable to complete self-administered questionnaires due to English language barrier, cognitive impairment, or severe medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the University of Washington Rhinology Clinic for evaluation of sinus problems
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg E Davis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States